CLINICAL TRIAL: NCT05021874
Title: The Effect of Different Physiotherapeutic Stimuli on Mandibular Analgesia and Range of Motion in Patients With Masticatory Muscles Disorder.
Brief Title: The Effect of Different Physiotherapeutic Stimuli on Stomatognathic System Structures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Dalewski Bartosz, DMD,PD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KB - 0012/102/13
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Pain; Stomatognathic Diseases; Muscle Hypertonia; Myofacial Pain Syndromes; Analgesia; Musculoskeletal Pain; Craniomandibular Osteopathy; Temporomandibular Disorder
Keywords: Pain; Physiotherapy; Range of motion; Temporomandibular Joint; Stomatognathic system
MeSH Terms: conditions — Pain; Stomatognathic Diseases; Muscle Hypertonia; Facial Neuralgia; Agnosia; Musculoskeletal Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physiotherapeutic procedures: magnetotherapy (Active Comparator): Magnetotherapy is a pulsating, non-homogeneous magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) will be applied using an elliptical applicator with a beam width of approx. 5 cm. Formative procedures within the masseter muscle, duration of the session amounted to 12 minutes. Physiotherapy treatment of the masseter muscles for a period of 10 days.
  Interventions: Other: Four different physiotherapy treatment
- Physiotherapeutic procedures:magneto-led therapy (Active Comparator): Magneto-led therapy is a synergistic action of a slowly changing magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) and LED diodes with the wavelength of 860 nm were applied using an elliptic magnetic-light (IR) applicator with a diameter of 5 [cm] containing 47 infrared diodes. Formative procedures within the masseter muscle, duration of the session amounted to 12 minutes. Physiotherapy treatment of the masseter muscles for a period of 10 days.
  Interventions: Other: Four different physiotherapy treatment
- Physiotherapeutic procedures:magneto-laser therapy (Active Comparator): Magneto-laser therapy is a synergistic action of a slowly changing magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) and a low-energy laser with infrared wavelength of 808 [nm] (max. power 300 mW) was applied. The dose was set to increase from 3,0 J/cm2 to 5,0 J/cm2 and the total dose applied per each patient from this subgroup was 40 J/cm2. Formative procedures within the masseter muscle, duration of the session amounted to 12 minutes. Physiotherapy treatment of the masseter muscles for a period of 10 days.
  Interventions: Other: Four different physiotherapy treatment
- Physiotherapeutic procedures: manual therapy of soft tissues (Active Comparator): Manual therapy of soft tissues will include: post-isometric relaxation of the masseter, cellular and tissue mobilization with Kibler fold, masseter trigger point therapy. Formative procedures within the masseter muscle, duration of the session amounted to 12 minutes. Physiotherapy treatment of the masseter muscles for a period of 10 days.
  Interventions: Other: Four different physiotherapy treatment

INTERVENTIONS:
Other: Four different physiotherapy treatment — Four different physiotherapy treatment will be used for, to reduce pain and tension in the masseter muscles. The assessment of pain intensity on the VAS scale will be assessed each time after the therapy. After the 10th day of therapy, it will be measured ROM.

SUMMARY:
The study will determinate influence of four selected physiotherapeutic procedures on the pain intensity and the range of mandibular mobility in patients with myofascial disorders in the SS.

DETAILED DESCRIPTION:
The study group will consist of 100 women (GI) aged 20 to 45 who report pain and increased facial muscle tension in masseter muscles.

The diagnosis will be made according to RDC/TMD (Research Diagnostic Criteria for Temporomandibular Disorders), which will determine the occurrence of painful myofascial disorders. Patients will undergo both external and intraoral dental examinations to exclude odontogenic and articular causes of pain. Patients will then be palpated for the masseter muscles and both: the range of mandibular abduction (linear measurement in mm) and the level of pain intensity (VAS scale).

The control group (GII) will consist of 100 women between 20 and 45 years of age with no signs of masticatory disorders or orofacial pain during a physical examination and with no such reference in their medical records.

In order to obtain a homogenic study group the following inclusion criteria will be applied:

* Myofascial pain of less than 12 months in duration that is evoked by an active motion of the mandible or by palpation.
* A feeling of an increased muscle tension
* Presence of all occlusal contact zones
* Female sex

Exclusion criteria:

* Past or present, neurological disease, neuromuscular disease or severe systemic disease.
* Temporomandibular joint pathology based on X-ray imaging or stomatological examination.
* Orthodontic or prosthetic treatment
* Contraindication to physiotherapeutic treatment

Patients with a stomatognathic system disorder will be randomized into four therapeutic subgroups, 26 patients each, who will receive a physiotherapy treatment of the masseter muscles for a period of 10 days (excluding Saturdays and Sundays). The duration of a single therapy session will be 12 minutes per patient in each of the subgroups.

The division of the study group into subgroups is as follows:

* IA: magnetotherapy; a pulsating, non-homogeneous magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) will be applied with an elliptical applicator with a beamwidth of approx. 5 cm.
* IB: magneto-led therapy; synergistic action of a slowly changing magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) and LED diodes with the wavelength of 860 nm will be applied with an elliptic magnetic-light (IR) applicator with a diameter of 5 [cm] containing 47 infrared diodes.
* IC: magneto-laser therapy; synergistic action of a slowly changing magnetic field generated by the Viofor JPS apparatus (Med & Life, Poland) and a low-energy laser with an infrared wavelength of 808 [nm] (max. power 300 mW) will be applied. The dose would increase from 3,0 J/cm2 to 5,0 J/cm2 and the total dose applied per each patient from this subgroup was 40 J/cm2.
* ID: manual therapy of soft tissues (i.e. post-isometric relaxation of the masseter, cellular and tissue mobilization with Kibler fold, masseter trigger point therapy).

Immediately after the therapy, the patients' pain level will be assessed via VAS scale. After the last day of physiotherapy, a linear measurement of mandibular abduction will be performed.

ELIGIBILITY:
Inclusion Criteria:

I. Myofacial pain of less than 12 months in duration that is evoked by an active motion of the mandible or by palpation.

II. Diagnosis according to RDC / TMD (Research Diagnostic Criteria for Temporomandibular Disorders), which showed painful myofascial disorders III. A feeling of an increased muscle tension IV. Presence of all occlusal contact zones V. Female sex

Exclusion Criteria:

I. Past or present, neurological disease, neuromuscular disease or a severe systemic disease.

II. Temporomandibular joint pathology based on X-ray imaging or stomatological examination.

III. Orthodontic or prosthetic treatment IV. Contraindication to physiotherapeutic treatment

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Famale
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 10 days
  Measurement on Visual Analogue Scale (VAS). It consists of a line, approximately 100 mm in length, at the left end of the scale "Score 0" witch means "no pain", at the right end of scale "Score 100mm" witch means "worst imaginable pain" [Time Frame: 10 days]
Measurement of the range of motion | 10 days
  Measurement of the range of mobility of the maximum abduction of the mandible (linear measurement from in mm. the upper to the lower incisor).
  [Time Frame: 10 days]

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Musculoskeletal System Rehabilitation, Pomeraniam Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gebska M, Dalewski B, Palka L, Kiczmer P, Kolodziej L. Kinesio Taping as an alternative therapy for limited mandibular mobility with pain in female patients with temporomandibular disorders: A randomized controlled trial. Dent Med Probl. 2024 Sep-Oct;61(5):659-670. doi: 10.17219/dmp/173126. PMID 38832764